CLINICAL TRIAL: NCT03262064
Title: Different Phenotypes of Bronchiectasis
Status: Terminated | Type: Observational
Why Stopped: Changing of specialty
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samah Mohammad Hussein, principal investigator, Assiut University
Other Study IDs: DPOB
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2017-09

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Pulmonary function tests,Bronchiectasis severity index score — Pulmonary function tests: including spirometry, DLCO, and lung volumes. Sputum investigations: The following investigations will be performed on fresh sputum samples; gram stains and culture, smear and culture for mycobacteria and fungi and antibiotic sensitivity tests Bronchoscopy: Bronchoscopy with bronchoalveolar lavage will be used to obtain specimens for staining and culture to identify type of colonization.
  Radiology: All patients will have a chest radiograph (PA and lateral) and high-resolution computed tomography (HRCT) scan.
  Bronchiectasis severity index score parameters FACED Score

SUMMARY:
Bronchiectasis is defined as abnormal chronic dilatation of one or more bronchi. Patients have a structural abnormality of the bronchial wall that predisposes them to bacterial infection likely due to impaired mucus clearance. A vicious cycle of chest infections and chronic lung inflammation can lead to further damage of the bronchial wall and spread of disease to normal areas of bystander lung.

DETAILED DESCRIPTION:
A search for an underlying cause, which may be amenable to a targeted intervention to prevent ongoing damage, is essential but often fruitless, and the focus of therapy rapidly turns to empiric treatments to prevent infective exacerbations and retard disease progression. The British Thoracic Society Bronchiectasis management guidelines provide an in-depth summary of the available literature and are an excellent tool for guiding treatment decision making. However, they do not provide guidance on which patients are most likely to benefit from specific interventions.Disease severity in bronchiectasis is hard to define. Radiological severity grading scores exist; however, there is often a disconnect between radiological severity, symptom burden and disease progressionIn 2014, competing bronchiectasis severity scores were published (FACED and the Bronchiectasis Severity Index (BSI).

In each of these, a combination of patient demographics, symptom scores, comorbidities, and clinical, radiological and microbiological parameters were used to construct scoring systems.

In case of the BSI, it predicted future mortality, and in the case of FACED, extended to prediction of future exacerbation frequency, hospitalisation and quality of life.These severity scores have utility in identifying an individual's risk of disease progression to a predefined outcome and aid in sub classifying this heterogeneous group of patients in a manner that may pave the way to future mechanistic studies, which explain how these different disease phenotypes arise and inform the development of targeted therapeutics.

ELIGIBILITY:
Inclusion Criteria:

patient diagnosed as bronchiectasis according to clinical picture and high- resolution computed tomography scan of the chest.

can perform pulmonary function test.

Exclusion Criteria:

No

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients (age >18and <70 years old) who will be presented to Assuit Chest Department from August 2017 till August 2018 and diagnosed as bronchiectasis according to clinical picture and high- resolution computed tomography scan of the chest.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
( Severity of Bronchiectasis will be measured according to BSI scoring system and FACED scoring system | Baseline
  BSI (Bronchiectasis severity index) score parameters include: Age, Body mass index, %FEV1 predicted, Previous Hospital admissions, Number of exacerbations in previous year, MRC dyspnea scale, Pseudomonas colonization, colonization with other organisms and radiological severity.
  Scoring:
  0-4 points Mild bronchiectasis 5-8points Moderate bronchiectasis 9+ points Severe bronchiectasis FACED score F - FEV1 A - Age C - Chronic colonization E - Radiological Extension D - Dyspnea
  Scoring:
  0-2 points Mild bronchiectasis 3-4 points Moderate bronchiectasis 5-7 points Severe bronchiectasis

SECONDARY OUTCOMES:
management of bronchectasis according to severity index | Baseline
  we will modify treatment of bronchectasis according to different phenotypes of bronchiectasis and severity score.

CONTACTS AND LOCATIONS:
Overall Officials: Maha El-kholy, Prof, Study Director
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Wilson CB, Jones PW, O'Leary CJ, Hansell DM, Cole PJ, Wilson R. Effect of sputum bacteriology on the quality of life of patients with bronchiectasis. Eur Respir J. 1997 Aug;10(8):1754-60. doi: 10.1183/09031936.97.10081754. PMID 9272915
- [Background] Eshed I, Minski I, Katz R, Jones PW, Priel IE. Bronchiectasis: correlation of high-resolution CT findings with health-related quality of life. Clin Radiol. 2007 Feb;62(2):152-9. doi: 10.1016/j.crad.2006.08.015. PMID 17207698
- [Background] Chalmers JD, Goeminne P, Aliberti S, McDonnell MJ, Lonni S, Davidson J, Poppelwell L, Salih W, Pesci A, Dupont LJ, Fardon TC, De Soyza A, Hill AT. The bronchiectasis severity index. An international derivation and validation study. Am J Respir Crit Care Med. 2014 Mar 1;189(5):576-85. doi: 10.1164/rccm.201309-1575OC. PMID 24328736
- [Background] Martinez-Garcia MA, de Gracia J, Vendrell Relat M, Giron RM, Maiz Carro L, de la Rosa Carrillo D, Olveira C. Multidimensional approach to non-cystic fibrosis bronchiectasis: the FACED score. Eur Respir J. 2014 May;43(5):1357-67. doi: 10.1183/09031936.00026313. Epub 2013 Nov 14. PMID 24232697